CLINICAL TRIAL: NCT07335718
Title: Evaluation of the Effectiveness of Focused Radiofrequency (TECAR) Therapy on Pain, Disability, Function, and Quality of Life in Patients With Lumbar Disc Herniation
Acronym: TECAR THERAPY
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Cemre Saymaz, DOCTOR, Ankara City Hospital Bilkent
Other Study IDs: TABED 1-24-833
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar Disc Herniation; TECAR Therapy; Pain
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TECAR Therapy: Patients with lumbar disc herniation
  Interventions: Device: TECAR THERAPY
- sham TECAR Therapy: Patients with lumbar disc herniation
  Interventions: Device: TECAR Therapy

INTERVENTIONS:
Device: TECAR THERAPY — TECAR therapy applied by a technician for 20 minutes per session, three days per week, for a total of six sessions
  Groups: TECAR Therapy
Device: TECAR Therapy — TECAR therapy is a new and effective treatment modality.
  Groups: sham TECAR Therapy

SUMMARY:
Low back pain is a very common health problem in societies, regardless of the underlying cause. Its lifetime prevalence has been reported to be as high as 75-80%. Low back pain negatively affects the quality of life of affected individuals. In addition to diagnostic and treatment costs, it can lead to serious physical disability, resulting in loss of workforce and placing a substantial economic burden on countries. Many different factors play a role in the etiology of low back pain. According to etiology, it can be classified as idiopathic, mechanical, rheumatologic, metabolic, endocrine, infectious, neoplastic, neurologic/psychiatric disorders, and pain of visceral origin. The treatment of low back pain can be classified into medical treatment, physical therapy, percutaneous invasive interventions, and surgical intervention. TECAR therapy is also one of the treatment modalities routinely used in clinical practice. Our aim is to develop more effective physical therapy programs.

DETAILED DESCRIPTION:
The study is planned as a prospective, randomized, double-blind trial. According to power analysis, 54 patients will be included to achieve 95% power. Eligible participants will be women or men aged 20-60 years who are diagnosed with lumbar disc herniation, have low back pain lasting longer than 12 weeks, present to the Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital as outpatients, and consent to participate in the study.

According to the study criteria, initial evaluations will be performed by a single Physical Medicine and Rehabilitation physician. Demographic data of eligible patients, including age, sex, height, weight, occupation, and systemic diseases, will be recorded.

Patients will be evaluated before treatment, immediately after treatment, and one month after the end of treatment using the following scales: Visual Analog Scale (VAS) for pain, Numeric Rating Scale (NRS), Quality of Life Scale (SF-36), Roland-Morris Disability Questionnaire, Oswestry Disability Index, Finger-to-Floor Distance Measurement, Beck Depression Inventory, and Lumbar Schober Test.

Patients will be divided into two groups. The first group will receive a home exercise program including lumbar active range of motion exercises and lumbar isometric strengthening exercises, performed five times per week for three weeks according to the level of movement restriction and pain severity, along with TECAR therapy applied by a technician for 20 minutes per session, three days per week, for a total of six sessions.

The second group will receive the same home exercise program-including lumbar active range of motion exercises and lumbar isometric strengthening exercises-performed five times per week for three weeks according to the level of movement restriction and pain severity, along with sham TECAR therapy applied by a technician for 20 minutes per session, three days per week, for a total of six sessions.

ELIGIBILITY:
Inclusion Criteria:

* Having low back pain lasting longer than 12 weeks

Having a diagnosis of lumbar disc herniation (bulging, protruded, or extruded)

Being able to comply with the exercise program

Willingness to participate in the study Being between 20 and 60 years of age

Exclusion Criteria:

Being younger than 20 years or older than 60 years

Having a known and/or newly diagnosed malignancy

Presence of cardiac implants such as a pacemaker

Having inflammatory low back pain

Having absolute spinal stenosis (anteroposterior diameter of the spinal canal < 10 mm and anteroposterior diameter of the lateral recess < 3 mm)

History of surgery due to lumbar disc herniation, lumbar spinal stenosis, vertebral fracture, or similar conditions

Presence of lumbar spondylolisthesis

Patients with sequestered disc herniation

Patients with polyneuropathy

Patients with central pain following stroke

Patients with neurological deficits

Having a diagnosed neurodegenerative disease

Having a systemic musculoskeletal disease

Patients with acute deep vein thrombosis

Pregnancy

Presence of infection at the skin surface where treatment will be applied

Unexplained weight loss

Bladder and/or bowel incontinence

Having received physical therapy modalities or injections for low back pain within the last 1 month

Having cognitive impairment

Refusal to participate in the study

-

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients presenting to the outpatient clinic of the Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Up to 1 month after the end of treatment
  Zero indicates no pain at all, whereas ten represents the most severe pain imaginable.

SECONDARY OUTCOMES:
Oswestry Disability Index | Up to 1 month after the end of treatment
  The Oswestry Disability Index (ODI) is a standardized questionnaire designed to assess the degree of disability and functional impairment in individuals with lower back pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I am undecided because the study is currently ongoing.